CLINICAL TRIAL: NCT02852096
Title: Assessing Her2/Neu Expression in Gastric Cancer With Dual or Multiple Tumor Tissue Paraffin Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: B2015-055R
Record Dates: First submitted 2015-11-08; First posted 2016-08-02 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Gastric Cancer; HER-2
Keywords: gastric cancer; Her2/neu; dual paraffin blocks; trastuzumab
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual or Multiple Paraffin Blocks (Experimental): Assessing Her2/neu Expression in Gastric Cancer with Dual or Multiple Tumor Tissue Paraffin Blocks
  Interventions: Other: Dual or Multiple Paraffin Blocks
- One Paraffin Blocks (Active Comparator): Assessing Her2/neu Expression in Gastric Cancer with One Tumor Tissue Paraffin Blocks
  Interventions: Other: One Paraffin Blocks

INTERVENTIONS:
Other: Dual or Multiple Paraffin Blocks — Assessing Her2/Neu Expression in Gastric Cancer With Dual or Multiple Tumor Tissue Paraffin Blocks
  Arms: Dual or Multiple Paraffin Blocks
Other: One Paraffin Blocks — Assessing Her2/Neu Expression in Gastric Cancer With One Tumor Tissue Paraffin Blocks
  Arms: One Paraffin Blocks

SUMMARY:
One paraffin block is routinely used for Human Epidermal Growth Factor Receptor 2 (Her2/neu) immunohistochemistry (IHC) assessment. Here, investigators investigated if picking two or multiple paraffin blocks for Her2/neu evaluation is an economical, efficient and practical method, which may reduce false-negativity of Her2/neu IHC assessment due to intratumoral heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 to 80; Received curative surgery with primary gastric adenocarcinoma; Did not receive any preoperative treatment.

Exclusion Criteria:

None.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The positive rate of cohort using dual or multiple tumor tissue paraffin blocks | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yingyong Hou, M.D. & Ph.D., Study Chair — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210